CLINICAL TRIAL: NCT06104462
Title: Exploring the Cortical Hemodynamic Variability of Prefrontal ITBS: a Concurrent TBS/fNIRS Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSEARS20220812002-02
Record Dates: First submitted 2023-10-20; First posted 2023-10-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cortical hemodynamic variability of iTBS and its courses (Experimental): A group of healthy adults shall undergo repeated experimental visits with concurrent TBS/fNIRS (3≤repetition≤15). An interval of at least two days (48 hours) between the visits is required to minimize carry-over effects from the iTBS protocols.
  Inter- (age, gender, personality inventory, etc.) and intra-individual factors (daily mood, daily sleep quality, physical activity levels, etc.) that are potentially moderating iTBS-induced excitability changes will be explored.
  Interventions: Device: Intermittent theta burst stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent theta burst stimulation (iTBS) — The iTBS protocol consists of 20 trains of stimulation. Each train comprises ten 3-pulse bursts, delivered at an intra-burst frequency of 50 Hz, with a 5 Hz overall frequency, followed by 8 seconds of rest. A total of 600 pulses (10*3*20) will be administered in this 3-minute iTBS protocol. Concurrent TBS/fNIRS stimulation will be applied over the left DLPFC at an intensity of 90% of the resting motor threshold (RMT), which is considered appropriate to ensure compliance and elicit robust DLPFC activation.
  Considering that the fNIRS optode beneath the coil increases the distance between the TMS coil and the skull by 10 mm, we will use the equation AdjMT% = MT + 2.8 * (Dsitex - Dm1). Therefore, 2.8 * 10 = 28% will be added to the normal intensity. The stimulation site over the DLPFC will be determined by the MNI coordinate (x-38, y+44, z+26) reported in previous studies.
  Other Names: Repetitive transcranial magnetic stimulation (rTMS)

SUMMARY:
An increasing number of studies have used the intermittent theta-burst stimulation (iTBS) protocol to investigate neural plasticity non-invasively in the prefontal cortex in healthy humans and in patients with psychiatric disorders. However, the variability in the neurophysiological response to iTBS stimulation is high. The cause of this variability is multifactorial and to some degree still unknown. Therefore, the current study explores inter- and intra-individual factors that are potentially moderating iTBS-induced excitability changes. A greater understanding of these determinants would be highly valuable for optimizing the therapeutic application of iTBS.

DETAILED DESCRIPTION:
The investigators will measure the cortical excitability induced by iTBS with concurrent TBS/fNIRS technique in the same healthy individuals on multiple testing days. Meanwhile, several potential inter- (age, gender, etc.) and intra-individual factors (daily mood, daily physical activity levels, etc.) recently identified in non-invasive transcranial brain stimulation studies will be assessed before applying iTBS to the same individual on each testing day.

ELIGIBILITY:
Inclusion Criteria:

* healthiness based on history and psychiatric assessment
* being able to hear and understand the verbal instructions
* completed at least 6 years of formal education

Exclusion Criteria:

* a current or past diagnosis of psychiatric, neurological disorders, or severe internal illness
* any conditions that will contraindicate to iTBS or fNIRS
* psychiatric disorders in their first-degree relatives
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Oxygenated hemoglobin (HbO) change compared to baseline | During and post TBS-fNIRS measurement, up to 3 months
  iTBS-induced HbO change in the DLPFC before, during and after stimulation

SECONDARY OUTCOMES:
Deoxygenated hemoglobin (HbR) change compared to baseline | During and post TBS-fNIRS measurement, up to 3 months
  iTBS-induced HbR change in the DLPFC before, during and after stimulation
Oxygen saturation change compared to baseline | During and post TBS-fNIRS measurement, up to 3 months
  iTBS-induced oxygen saturation change in the DLPFC before, during and after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Georg Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request
Access Criteria: Upon request